CLINICAL TRIAL: NCT04251026
Title: A Phase 1/2, Multicenter, Open-Label Study to Determine the Safety, Pharmacokinetics, and Pharmacodynamics of DNL310 in Pediatric Participants With Hunter Syndrome
Brief Title: A Study of Tividenofusp Alfa (DNL310) in Pediatric Participants With Hunter Syndrome
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Denali Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DNLI-E-0002; 2023-508619-22-00 (EU CTIS Number); 2019-004909-27 (EudraCT Number)
Record Dates: First submitted 2020-01-28; First posted 2020-01-31 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Mucopolysaccharidosis II
Keywords: MPS II; Hunter Syndrome; nMPS II
MeSH Terms: conditions — Mucopolysaccharidosis II; Sudden Infant Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Cohort A (Experimental): Dose escalation followed by a consistent dose level in participants with neuronopathic MPS II
  Interventions: Drug: tividenofusp alfa
- Cohort B (Experimental): A consistent dose level in participants with non-neuronopathic MPS II, neuronopathic MPS II, or unknown phenotype followed by dose escalation in some participants.
  Interventions: Drug: tividenofusp alfa
- Cohort C (Experimental): A consistent dose level in participants with neuronopathic MPS II
  Interventions: Drug: tividenofusp alfa
- Cohort D (Experimental): A consistent dose level in participants with non-neuronopathic MPS II or neuronopathic MPS II
  Interventions: Drug: tividenofusp alfa
- Cohort E (Experimental): A consistent dose level in participants with non-neuronopathic MPS II or neuronopathic MPS II
  Interventions: Drug: tividenofusp alfa

INTERVENTIONS:
Drug: tividenofusp alfa — Intravenous repeating dose

SUMMARY:
This is a multicenter, multiregional, open-label study to assess the safety, pharmacokinetics (PK), and pharmacodynamics (PD) of tividenofusp alfa (DNL310), an investigational central nervous system (CNS)-penetrant enzyme replacement therapy (ERT), designed to treat both the peripheral and CNS manifestations of Mucopolysaccharidosis type II (MPS II; Hunter syndrome).

Participants, whose physicians feel they are deriving benefit, will have the opportunity to be reconsented into a safety extension and then an open-label extension for continued evaluation.

ELIGIBILITY:
Key Inclusion Criteria:

* Confirmed diagnosis of MPS II
* Cohort A: Participants aged ≥5 to ≤10 years with neuronopathic MPS II
* Cohort B: Participants aged ≥1 to ≤18 years with non-neuronopathic MPS II, neuronopathic MPS II, or unknown phenotype
* Cohort C: Participants aged <4 years with neuronopathic MPS II (this cohort can include participants ≥4 to ≤18 years of age if participant is a blood relative of a participant <4 years of age)
* Cohort D: Participants aged ≤18 years with non-neuronopathic MPS II or neuronopathic MPS II with preexisting hepatomegaly who have never taken standard-of-care ERT
* Cohort E: neuronopathic MPS II participants aged ≥6 years at screening, non-neuronopathic MPS II participants <6 or ≥17 years at screening, and neuronopathic MPS II participants ≥1 to ≤18 years at screening with a history of prior haematopoietic stem cell transplantation or gene therapy who have completed at least 48 weeks in Study DNLI-E-0001
* For participants receiving intravenous iduronate 2-sulfatase (IDS) ERT, tolerated a minimum of 4 months of therapy during the period immediately prior to screening.

Key Exclusion Criteria:

* Unstable or poorly controlled medical condition(s) or significant medical or psychological comorbidity or comorbidities that, in the opinion of the investigator, would interfere with safe participation in the trial or interpretation of study assessments
* Use of any CNS-targeted MPS II ERT within 3 months before study start for participants aged ≥5 years, and within 6 months before study start for participants aged <5 years
* Use of IDS gene therapy or stem cell therapy at any time (except for participants in Cohort E)
* Clinically significant thrombocytopenia, other clinically significant coagulation abnormality, or significant active bleeding, or required treatment with an anticoagulant or more than two antiplatelet agents
* Contraindication for lumbar punctures
* Have a clinically significant history of stroke, status epilepticus, head trauma with loss of consciousness, or any CNS disease that is not MPS II-related within 1 year of screening
* Have had a ventriculoperitoneal (VP) shunt placed, or any other brain surgery, or have a clinically significant VP shunt malfunction within 30 days of screening
* Have any clinically significant CNS trauma or disorder that, in the opinion of the investigator, may interfere with assessment of study endpoints or make participation in the study unsafe

Max Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 47 (Actual)
Dates: Start 2020-07-16 (Actual); Primary Completion 2031-02 (Estimated); Study Completion 2031-02 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events (TEAEs) | 24 weeks, 104 weeks, and 357 weeks
Change from baseline in urine total glycosaminoglycan (GAG) concentrations | 24 weeks, 104 weeks, and 357 weeks
Incidence and severity of infusion-related reactions (IRRs) | 24 weeks, 104 weeks, and 357 weeks
Change from baseline in concomitant medications | 24 weeks, 104 weeks, and 357 weeks

SECONDARY OUTCOMES:
Percentage change from baseline in cerebrospinal fluid (CSF) of heparan sulfate | 24 weeks
Participants with improvement in individual disease progression in the Vineland Adaptive Behavior Scale Adaptive Behavior Composite (ABC) score | 49 weeks
Participants with improvement in individual disease progression in the Vineland Adaptive Behavior Scale subdomain scores | 49 weeks
PK parameter: Maximum observed concentration (Cmax) of DNL310 in serum | 24 weeks
PK parameter: Trough concentration (Cmin) of DNL310 in serum | 24 weeks
PK parameter: Time to maximum observed concentration (tmax) of DNL310 in serum | 24 weeks
PK parameter: Area under the concentration-time curve from time zero to the time of last quantifiable concentration (AUClast) of DNL310 in serum | 24 weeks
PK parameter: Area under the concentration-time curve from time zero to infinity (AUC∞) of DNL310 in serum | 24 weeks
PK parameter: Area under the concentration-time curve over a dosing interval (AUCτ) of DNL310 in serum | 24 weeks
PK parameter: Apparent terminal elimination half-life (t½) of DNL310 in serum | 24 weeks
Characterization of immunogenicity of DNL310 in serum, as measured by the incidence of anti-drug antibodies (ADAs) relative to baseline | 24 weeks
Percent change from baseline in urine concentration of heparan sulfate (HS) | 24 weeks
Participants with liver volume in the normal range | 24 weeks and 49 weeks
Percentage change from baseline in liver volume | 24 weeks and 49 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sam Lu, MD, Study Director — Denali Therapeutics
Locations (7):
- United States (4):
  - UCSF Benioff Children's Hospital, Oakland, California
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - UNC Children's Research Institute, Chapel Hill, North Carolina
  - UPMC | Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
- McGill University Health Centre - Royal Victoria Hospital, Montreal, Quebec, Canada
- Erasmus Medical Center, Rotterdam, South Holland, Netherlands
- St Mary's Hospital, Manchester Academic Health Science Centre, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Muenzer J, Burton BK, Harmatz P, Rajan DS, Jones SA, van den Hout JMP, Mitchell JJ, Bhalla A, Engmann NJ, Zubizarreta I, Dong W, Model F, Watts RJ, Troyer MD, Chin PS, Ho C. An Intravenous Brain-Penetrant Enzyme Therapy for Mucopolysaccharidosis II. N Engl J Med. 2026 Jan 1;394(1):39-50. doi: 10.1056/NEJMoa2508681. PMID 41467650